CLINICAL TRIAL: NCT05172219
Title: A Quality Improvement Randomized Clinical Trial to Evaluate Electronic Portal Messaging, Embedded Asynchronous Care and Physician Versus System as Message Sender on Physician-Assisted Smoking Quit Attempts of Primary Care, Adult Patients
Brief Title: Evaluation of Electronic Portal Messaging and Embedded Asynchronous Care on Physician-Assisted Smoking Quit Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2020031
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Smoking, Tobacco
Keywords: Smoking Quit Attempts; Quality Improvement; Asynchronous Care; Electronic Messaging
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: The model was a 2 (link to survey) × 2 (message source) experimental design; therefore, we had two factors that created four treatment conditions.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants: The patients were not informed of other portal messages. The portal message they received (if it had a link to asynchronous care or not and if it was sent by physician or system) was determined by random assignment.
  Care Providers: After reviewing patients for exclusion criteria, the physicians were not informed which intervention group patients were assigned. They knew who was selected for the study and then those patients were randomly assigned to intervention groups by computerized randomization system.
  Investigators: The data was extracted from the EHR and de-identified prior to sharing it with the investigators. Therefore, the investigators were blind to patients and patient assignment.
  Outcomes Assessor: Outcomes were assessed only from de-identified data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Message Type PNSL: Physician sender, No Survey Link (Active Comparator): In this arm, the Physician is message sender and the message does not include a link to a survey that initiates asynchronous care.
  Interventions: Behavioral: Physician Sent Outreach without Embedded Asynchronous Care in Portal Message
- Message Type PSL: Physician sender, Survey Link (Active Comparator): In this arm, the Physician is message sender and the message does include a link to a survey that initiates asynchronous care.
  Interventions: Behavioral: Physician Sent Outreach with Embedded Asynchronous Care in Portal Message
- Message Type SNSL: System sender, No Survey Link (Active Comparator): In this arm, the Health System is message sender and the message does not include a link to a survey that initiates asynchronous care.
  Interventions: Behavioral: System Sent Outreach without Embedded Asynchronous Care in Portal Message
- Message Type SSL: System sender, Survey Link (Active Comparator): In this arm, the Health System is message sender and the message does include a link to a survey that initiates asynchronous care.
  Interventions: Behavioral: System Sent Outreach with Embedded Asynchronous Care in Portal Message

INTERVENTIONS:
Behavioral: Physician Sent Outreach with Embedded Asynchronous Care in Portal Message — PCPs sent a portal message encouraging a quit attempt embedded a link to asynchronous care within a portal message encouraging a quit attempt in order to compare EMR-documented, physician-assisted quit attempts to those who received messages without the link 30 days after messages were sent.
  Other Names: PSL
  Arms: Message Type PSL: Physician sender, Survey Link
Behavioral: Physician Sent Outreach without Embedded Asynchronous Care in Portal Message — Physician sent a portal message encouraging a quit attempt without a link to asynchronous care within a portal message encouraging a quit attempt in order to compare EMR-documented, physician-assisted quit attempts to those who received messages without the link 30 days after messages were sent.
  Other Names: PNSL
  Arms: Message Type PNSL: Physician sender, No Survey Link
Behavioral: System Sent Outreach with Embedded Asynchronous Care in Portal Message — Health System sent a portal message encouraging a quit attempt embedded a link to asynchronous care within a portal message encouraging a quit attempt in order to compare EMR-documented, physician-assisted quit attempts to those who received messages without the link 30 days after messages were sent.
  Other Names: SSL
  Arms: Message Type SSL: System sender, Survey Link
Behavioral: System Sent Outreach without Embedded Asynchronous Care in Portal Message — Health System sent a portal message encouraging a quit attempt without a link to asynchronous care within a portal message encouraging a quit attempt in order to compare EMR-documented, physician-assisted quit attempts to those who received messages without the link 30 days after messages were sent. Half of the messages came from the patient's PCP and the other half came from the health system to determine if communication from a patient's physician was associated with more quit attempts.
  Other Names: SNSL
  Arms: Message Type SNSL: System sender, No Survey Link

SUMMARY:
Among 10 PCPs, 200 adult smokers with an active patient portal who had been seen by a PCP within 12 months were randomly selected and randomly assigned to one of four conditions to compare the quit attempts of patients sent electronic outreach with and without asynchronous care link and to compare the quit attempts of patients who recieved the portal message from PCP or the health system.

DETAILED DESCRIPTION:
The investigators compared the effects of four technology-based smoking cessation messaging strategies on quit attempts by smokers identified in the health system. Specifically, investigators used a fully crossed between-subjects 2 (link to survey on smoking cessation guide: yes/no) × 2 (message source: PCP-generated vs. health system-generated) experimental design to which participants were randomly assigned to one of four intervention groups using a computerized random number generator:

* Group 1 was sent the message from their physician without a link to a survey;
* Group 2 was sent the message from their physician with the link to the survey (which constitutes the asynchronous care);
* Group 3 was sent the message from the health system without a link to the survey; and
* Group 4 was sent the message from the health system with the link to the survey (which constitutes the asynchronous care).

Electronic outreach was a message sent to patients via the patient portal. It encouraged a quit attempt; offered physician assistance; advised the patient on medication use to control cravings; and offered counseling support in the form of a Quitline. Patients in Groups 1 and 3 were invited to schedule an in-person appointment with their PCP if they wanted help. Patients in Groups 2 and 4 received the message with an embedded link to Tobacco Cessation Survey to receive PCP assistance asynchronously. If patients clicked through to access the survey, they answered 17 questions, confirming smoking status, reporting safety information for medication selection, describing prior quit attempts and sharing treatment preferences. The intervention was "asynchronous" because it did not involve direct, simultaneous interaction (e.g., face-to-face, chat, video conference) between the physician and the patient. After patient responses were submitted, they were stored and forwarded to their PCP. Physicians communicated the care plan and instructed patients via the portal message. If the plan included medication, a prescription was sent to the patient's EHR-documented preferred pharmacy without an in-person visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older who were designated as a smoker in the EHR who had at least one face-to-face visit with their PCP in the prior 12 months and had a patient portal account
* To ensure equal representation across the 10 physicians, we randomly selected 20 patients under each physician to serve in the sample.

Exclusion Criteria:

* Patients were excluded if they no longer see the PCP, had a diagnosis for which the outreach program would be insensitive (e.g., lung cancer), previously expressed not wanting smoking cessation counseling, or were no longer a smoker.
* (Patients were post-hoc excluded if EHR indicated that they had received smoking cessation treatment 60 days prior to portal message intervention.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Smoking Quit Attempt | 30 days after intervention
  Smoking Quit Attempt documented in the EMR

OTHER OUTCOMES:
Physician Perceptions of Electronic Outreach Intervention | 6 months after intervention
  Physician perceptions of the electronic outreach intervention were measured using a 5-point scale to assess perceptions of workload, comfort of providing medication from survey information, and further interest in the program.

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie A Erdmann, MS, Principal Investigator — Oklahoma State University
Locations (1):
- Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erdmann M, Edwards B, Adewumi MT. Effect of Electronic Portal Messaging With Embedded Asynchronous Care on Physician-Assisted Smoking Cessation Attempts: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220348. doi: 10.1001/jamanetworkopen.2022.0348. PMID 35226082